CLINICAL TRIAL: NCT03179085
Title: Home-Based Chronic Kidney Disease (CKD) Care in Native American's of New Mexico- A Disruptive Innovation
Brief Title: Home-Based Kidney Care in Native American's of New Mexico (HBKC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Vallabh O Shah, Professor, University of New Mexico
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-344
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Diabetes; American Indians; Disparity; microalbuminuria; Telemedicine; Community health representative (CHR); Patient Activation Measure (PAM); Home base kidney care
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants randomized to control group will receive standard care for 12 months before entering into the delayed intervention. Participants randomized to the intervention will receive the intervention during the first 12 months.
  We want to clarify that a total of 529 individuals were consented for participation in the study. These participants responded to screening questionnaires which included POC testing, Blood pressure, medical history and physical assessments. From those 529 participants, a total of 286 did not meet inclusion criteria for randomization and 57 declined further participation in the study. Therefore, we randomized 186 participants, 93 to the HBKC care intervention and 93 to the Delay Intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care / Delayed Intervention (Active Comparator): Participants randomized to the control group will receive usual care by their provider for 12 months. They will also attend one group class taught by CHRs in which they will learn basic information about diabetes prevention. DI participants will receive publicly-available literature that reinforces the information given in class, and they will have no other contact with study staff aside from during study data collection visits at baseline and 12 months. After 12 months of usual care, patients will enter into the delayed intervention where they will complete 12 months of Home-Based Kidney Care (HBKC).
  Interventions: Behavioral: Home-Based Kidney Care
- Home-Based Kidney Care Intervention (Experimental): All subjects randomized to the HBKC arm will be visited by a CHR in their home at least every two weeks for the duration of the 12 month intervention. Each visit will last 30 minutes to one hour and participant preference will be incorporated into the HBKC intervention arm by allowing participants to prioritize the order in which curriculum topic areas will be emphasized by the CHRs. Topics from currently available NIDDK and IHS kidney education materials will include: (1) Kidney 101, (2) weight management, (3) exercise, (4) healthy eating, (5) medication management, (6) coping with stress, (7) risk factor management (i.e.- blood pressure, hyperlipidemia), (8) alcohol and substance abuse, (9) smoking cessation, and related health concerns.
  Interventions: Behavioral: Home-Based Kidney Care

INTERVENTIONS:
Behavioral: Home-Based Kidney Care — All subjects randomized to the HBKC arm will be visited by a community health representative in their home at least every two weeks for the duration of the 12 month intervention. Each visit will last 30 minutes to one hour and cover materials like, (1) Kidney 101, (2) weight management, (3) exercise, (4) healthy eating, (5) medication management, (6) coping with stress, (7) risk factor management (i.e.- blood pressure, hyperlipidemia), (8) alcohol and substance abuse, (9) smoking cessation, and related health concerns.

SUMMARY:
People reach End Stage Renal Disease (ESRD) due to progressive chronic kidney disease (CKD). CKD is associated with increased risk for heart disease and death. The burden of chronic kidney disease is increased among minority populations compared to Caucasians. New Mexico American Indians are experiencing an epidemic of chronic kidney disease due primarily to the high rates of obesity and diabetes. The present study entitled Home-Based Kidney Care is designed to delay / reduce rates of ESRD by early interventions in CKD. Investigators propose to assess the safety and efficacy of conducting a full-scale study to determine if home based care delivered by a collaborative team composed of community health workers, the Albuquerque Area Indian Health Board and University of New Mexico faculty will decrease the risk for the development and the progression of CKD.

DETAILED DESCRIPTION:
Hypothesis:

Specific Aim 1: Screen 600 participants from four different American Indian tribes in New Mexico to identify incident cases of CKD and identify participants for the proposed study of HBKC;

Specific Aim 2: Conduct a 12 month study of HBKC among 240 Native Americans randomized in a 1:1 allocation to HBKC group versus Delayed Intervention (DI) group to demonstrate improvement in Patient Activation Measures (PAM) and adherence to treatment. We will demonstrate that CKD clinical risk profiles will improve with HBKC as compared to DI at 12 months and 4 months post intervention (16 months);

Specific Aim 3: To demonstrate that HBKC will improve psychological factors that map onto important cultural variations in treatment efficacy and health outcomes. Specifically, we will show improvement in potential mediators (treatment engagement, self-efficacy, coping and increased knowledge) and moderators (stigma, and chronic stress, and depression) of health disparity and outcome.

Study Outcomes: (1) The patient activation measures and adherence; (2) Changes in clinical phenotypes including Cr, UACR, A1c, body weight, BMI, fasting glucose, blood pressure (BP), plasma lipids, and inflammatory markers; (3) Changes in the quantitative traits such as diet and scores from a battery of mental-health, self-efficacy, and quality of life instruments.

Health Impact: The active participation of New Mexico tribal leadership and the Albuquerque Area Indian Health Board, as well as the accessibility to native CHR personnel, render the outcomes that will be demonstrated by this proposal easily sustainable over the long term. If successful, this program has the potential to change best-practices for CKD progression and to reduce health disparities in a cost-effective and sustainable manner.

ELIGIBILITY:
Inclusion Criteria:

* (1) live in a household with 1 participant
* (2) age 21 to 80 years
* (3) negative pregnancy test in women of child-bearing potential
* (4) diagnosed diabetics or HbA1c >7
* (5) BMI >27 kg/m2 and UACR of >/= 30

Exclusion Criteria:

* (1) life expectancy < 1 year
* (2) pregnancy or absence of reliable birth control in women of child-bearing potential
* (3) malignancy except non-melanoma skin cancer
* (4) blind
* (5) ESRD and on dialysis
* (6) kidney transplant recipient
* (7) unwilling or unable to give informed consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vallabh Shah, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be available to share once the tribal leadership approves it.

REFERENCES:
- [Background] Cukor D, Cohen LM, Cope EL, Ghahramani N, Hedayati SS, Hynes DM, Shah VO, Tentori F, Unruh M, Bobelu J, Cohen S, Dember LM, Faber T, Fischer MJ, Gallardo R, Germain MJ, Ghahate D, Grote N, Hartwell L, Heagerty P, Kimmel PL, Kutner N, Lawson S, Marr L, Nelson RG, Porter AC, Sandy P, Struminger BB, Subramanian L, Weisbord S, Young B, Mehrotra R. Patient and Other Stakeholder Engagement in Patient-Centered Outcomes Research Institute Funded Studies of Patients with Kidney Diseases. Clin J Am Soc Nephrol. 2016 Sep 7;11(9):1703-1712. doi: 10.2215/CJN.09780915. Epub 2016 May 19. PMID 27197911
- [Background] Shah VO, Carroll C, Mals R, Ghahate D, Bobelu J, Sandy P, Colleran K, Schrader R, Faber T, Burge MR. A Home-Based Educational Intervention Improves Patient Activation Measures and Diabetes Health Indicators among Zuni Indians. PLoS One. 2015 May 8;10(5):e0125820. doi: 10.1371/journal.pone.0125820. eCollection 2015. PMID 25954817
- [Background] Newman S, Cheng T, Ghahate DM, Bobelu J, Sandy P, Faber T, Shah VO. Assessing knowledge and attitudes of diabetes in Zuni Indians using a culture-centered approach. PLoS One. 2014 Jun 11;9(6):e99614. doi: 10.1371/journal.pone.0099614. eCollection 2014. PMID 24919064
- [Background] Shah VO, Ghahate DM, Bobelu J, Sandy P, Newman S, Helitzer DL, Faber T, Zager P. Identifying barriers to healthcare to reduce health disparity in Zuni Indians using focus group conducted by community health workers. Clin Transl Sci. 2014 Feb;7(1):6-11. doi: 10.1111/cts.12127. Epub 2013 Nov 8. PMID 24528897
- [Background] MacCluer JW, Scavini M, Shah VO, Cole SA, Laston SL, Voruganti VS, Paine SS, Eaton AJ, Comuzzie AG, Tentori F, Pathak DR, Bobelu A, Bobelu J, Ghahate D, Waikaniwa M, Zager PG. Heritability of measures of kidney disease among Zuni Indians: the Zuni Kidney Project. Am J Kidney Dis. 2010 Aug;56(2):289-302. doi: 10.1053/j.ajkd.2010.03.012. Epub 2010 Jun 19. PMID 20646805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 529 individuals were consented for participation in the study. These participants responded to screening questionnaires which included POC testing, Blood pressure, medical history and physical assessments. From those 529 participants, a total of 286 did not meet inclusion criteria for randomization and 57 declined further participation in the study. Therefore, we randomized 186 participants, 93 to the HBKC care intervention and 93 to the Delay Intervention.
Pre-assignment Details: The study enrolled males and females who displayed evidence of diabetic chronic kidney disease and who: were age 21 to 80 years; had a negative pregnancy test in women of child-bearing potential; were diagnosed diabetics or HbA1c >7; had BMI >27 kg/m2, and had UACR >=30 mg/g. Exclusion criteria: life expectancy < 1 year; absence of reliable birth control in women of child-bearing potential; malignancy except non-melanoma skin cancer; blind; and unwilling or unable to give informed consent.
Period: Overall Study
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Started | 93 | 93
Completed | 93 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention | Total
Number analyzed (Participants) | 93 | 93 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing age data for some participants.
  years
    number analyzed (Participants) | 91 | 92 | 183
    (all) | 57.2 (14.8) | 56.1 (14.6) | 56.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing gender data for some participants.
  Participants
    number analyzed (Participants) | 92 | 92 | 184
    Female | 52 | 52 | 104
    Male | 40 | 40 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 93 | 93 | 186
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Patient Activation Measure (PAM)
Description: Assesses an individual's knowledge, skill, and confidence for managing one's health and healthcare. PAM total scores have a theoretical range from 0 to 100, with higher scores representing greater patient activation.
Time Frame: Baseline, 6 and 12 months
Population: Missing PAM scores data and the number differ for each time point. Participants were invited to participate at each time point regardless of participation in other study periods. We note that this study took place during COVID 19 pandemic.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 92 | 92
score on a scale
  Baseline PAM scores: number analyzed (Participants) | 77 | 86
  Baseline PAM scores | 60.8 (2.12) | 61.5 (2.06)
  6-month change in PAM scores: number analyzed (Participants) | 23 | 53
  6-month change in PAM scores | 1.73 (1.64) | 3.44 (1.55)
  12-month change in PAM scores: number analyzed (Participants) | 33 | 37
  12-month change in PAM scores | 2.28 (2.05) | 3.59 (1.94)

2. Secondary Outcome: HbA1c
Description: Hemoglobin A1C measured as percent of glycosylated high hemoglobin cells
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Not all enrolled participants provided a baseline blood sample which resulted in fewer analyzed than enrolled.
Measure: Mean (Standard Deviation); unit: percent of cells
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 65 | 72
percent of cells
  Baseline | 8.65 (2.13) | 8.54 (2.25)
  Change from baseline to 6 months: number analyzed (Participants) | 29 | 45
  Change from baseline to 6 months | -0.31 (2.80) | -0.34 (1.97)
  Change from baseline to 12 months: number analyzed (Participants) | 23 | 35
  Change from baseline to 12 months | -0.23 (1.74) | -0.18 (2.14)

3. Secondary Outcome: Blood Glucose Levels
Description: amount of glucose in the blood measured as mg/dL - milligrams per deciliter
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Analysis were restricted to those who provided valid blood samples.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 65 | 73
milligrams per deciliter
  Baseline | 172.06 (87.12) | 183.18 (111.64)
  Change from baseline to 6months: number analyzed (Participants) | 31 | 46
  Change from baseline to 6months | 24.06 (103.02) | -10.59 (100.03)
  Change from baseline to 12 months: number analyzed (Participants) | 26 | 35
  Change from baseline to 12 months | 28.62 (79.19) | 3.26 (110.88)

4. Secondary Outcome: HDL
Description: High density lipoprotein as mg/dL - milligrams per deciliter
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Analysis were restricted to those who provided valid blood samples.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 65 | 71
milligrams per deciliter
  Baseline | 46.08 (12.58) | 46.38 (12.03)
  Change from baseline to 6 months: number analyzed (Participants) | 29 | 41
  Change from baseline to 6 months | 0.21 (6.93) | -0.61 (7.25)
  Change from baseline to 12 months: number analyzed (Participants) | 23 | 34
  Change from baseline to 12 months | -1.83 (7.95) | -1.59 (8.94)

5. Secondary Outcome: LDL
Description: Low density lipoprotein as mg/dL - milligrams per deciliter
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Analysis were restricted to those who provided valid blood samples.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 64 | 69
milligrams per deciliter
  Baseline | 73.66 (31.59) | 77.54 (48.11)
  Change from baseline to 6 months: number analyzed (Participants) | 29 | 39
  Change from baseline to 6 months | 12.59 (72.37) | -8.33 (48.49)
  Change from baseline to 12 months: number analyzed (Participants) | 22 | 31
  Change from baseline to 12 months | 4.18 (23.08) | 11.81 (25.00)

6. Secondary Outcome: Creatinine
Description: Serum creatinine measured as mg/dL - milligrams per deciliter
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Analysis were restricted to those who provided valid blood samples.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 65 | 73
milligrams per deciliter
  Baseline | 0.78 (0.27) | 0.80 (0.34)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 46
  Change from baseline to 6 months | 0.10 (0.31) | 0.14 (0.51)
  Change from baseline to 12 months: number analyzed (Participants) | 26 | 36
  Change from baseline to 12 months | 0.03 (0.19) | 0.21 (0.59)

7. Secondary Outcome: SF12 Physical
Description: KDQOL Short Form 12 (SF12) Physical functioning T score: normal mean=50, normal standard deviation=10. Higher values is higher quality of life.
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Analysis were restricted to those who completed the KDQOL instrument.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 73 | 78
T score
  Baseline | 43.50 (9.88) | 44.43 (8.02)
  Change from baseline to 6 months: number analyzed (Participants) | 21 | 38
  Change from baseline to 6 months | -2.07 (9.44) | -0.09 (8.43)
  Change from baseline to 12 months: number analyzed (Participants) | 17 | 32
  Change from baseline to 12 months | -1.18 (8.02) | -1.19 (9.39)

8. Secondary Outcome: SF12 Mental
Description: KDQOL Short Form 12 (SF12) Mental functioning T score: normal mean=50, normal standard deviation=10. Higher values is higher quality of life.
Time Frame: Baseline. Change from baseline at 6 and 12 months
Population: Analysis were restricted to those completed the KDQOL instrument
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
Number analyzed (Participants) | 73 | 78
T score
  Baseline | 50.42 (10.90) | 51.33 (9.68)
  Change from baseline to 6 months: number analyzed (Participants) | 21 | 38
  Change from baseline to 6 months | 1.96 (9.74) | 0.47 (11.94)
  Change from baseline to 12 months: number analyzed (Participants) | 17 | 32
  Change from baseline to 12 months | 4.56 (9.88) | 2.53 (11.84)

ADVERSE EVENTS:
Time Frame: There were no adverse events reported during the 12 month duration of the study.
Arm/Group | Usual Care / Delayed Intervention | Home-Based Kidney Care Intervention
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 0/93 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03179085/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03179085/SAP_001.pdf
  • Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03179085/ICF_002.pdf